CLINICAL TRIAL: NCT04253990
Title: Comparison Between EMR and Precut-EMR for Colorectal Polyp; Randomized Prospective Study
Brief Title: Efficacy and Safety of Precut-EMR for Resecting of Colonic Polyp
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dong-Hoon Yang, Clinical Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2015-1496-0001
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Colonic Polyps
Keywords: Colonic polyps; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precut-EMR (Experimental): For treating of 10~20mm colon polyp, patient will be randomly divided into two groups, a Precut-EMR group and a EMR group.
  In Precut-EMR, endoscopist submucosally inject with saline around a polyp. Subsequently, circumferential incision/precutting was made with the tip of the snare around 2 mm outside the tumor. After that, the snare was positioned in the cut groove and tightend, and the tumor was resected using electrical current.
  Interventions: Procedure: Precut EMR
- Conventional EMR (Active Comparator): For treating of 10~20mm colon polyp, patient will be randomly divided into two groups, a Precut-EMR group and a EMR group.
  Conventional EMR had been widely used technique. Endoscopist submucosally inject with saline around a polyp. After that, snare is positioned around a polyp, and polyp was resected using electrical current
  Interventions: Procedure: Conventional MER

INTERVENTIONS:
Procedure: Precut EMR — For treating of 10~20mm colon polyp, patient will be randomly divided into two groups, a Precut-EMR group and a EMR group.
  In Precut-EMR, endoscopist submucosally inject with saline around a polyp. Subsequently, circumferential incision/precutting was made with the tip of the snare around 2 mm outside the tumor. After that, the snare was positioned in the cut groove and tightend, and the tumor was resected using electrical current.
  Arms: Precut-EMR
Procedure: Conventional MER — EMR had been widely used technique. Endoscopist submucosally inject with saline around a polyp. After that, snare is positioned around a polyp, and polyp was resected using electrical current.
  Arms: Conventional EMR

SUMMARY:
This study was attempted to determine the efficacy and complication of precut EMR comparing with convetional EMR for resecting of 10 ~ 20 mm colon polyp through prospective, randomized controlled trial.

DETAILED DESCRIPTION:
In general, a potential risk of advanced colorectal neoplasia is proportional with size. However, recent study report that occurence rate of advanced neoplasia in small polyp is 9 ~ 10 %. And, incidence of interval cancer after screening colonoscopy was reported as 10 ~ 27%. So We can suspect that complete resection of small polyp is important. Previous study recommended that endoscopic submucosal dissection (ESD) is a safe and effective procedure for treating colon polyp larger than 20 mm because of high complete resection rate and low recurrence rate. In contrast, endoscopic mucosal resection (EMR) is more recommended for resecting colon polyp smaller than 20 mm because of technical ease and low rate of complication.

However, Complete resection rate of conventional EMR is 60 ~ 70%. In case of incomplete resection, local recurrence rate is higher than complete resection. And In case of adenocarcinoma, specimen of piecemeal resection cannot be evaluated a depth of invasion and resection margin, and physician cannot decide a therapeutic plan.

In precut-EMR, mucosal resection is performed after pre-incision around a polyp. When precut EMR of polyp > 20 mm was performed in previous study, complete resection rate and en-bloc resection rate were higher and local recurrence rate was lower than conventional EMR. But, there is no study of comparsion precut EMR and conventional EMR for resecting colon polyp < 20 mm. This study was attempted to determine the efficacy and complication of precut EMR comparing with convetional EMR through prospective, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 20 years old who had 10~20 mm colon polyp and agreed to participate a research

Exclusion Criteria:

* Medication history of antiplatelet agent within a week of procedure.
* Medical history of coagulopathy
* More than American Society of Anesthesiology class III
* Medical history of liver cirrhosis, chronic kidney disease, malignancy, inflammatory bowel disease, severe inflammatory disease.
* pedunculated polyp and polyp with malignant potential.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Histologic complete resection rate | baseline ( enrollment of all planned patient)

SECONDARY OUTCOMES:
Procedure time | procedure
Complication such as perforation, bleeding | baseline ( enrollment of all planned patient)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-hoon Yang, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No